CLINICAL TRIAL: NCT04872127
Title: Distal Versus Proximal Protection on Cerebral Microembolization During High-risk Carotid Artery Stenting
Acronym: MOSCASH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: device unavailable
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: MOSCASH
Record Dates: First submitted 2021-04-30; First posted 2021-05-04 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Stroke; Carotid Stenosis
Keywords: carotid stenting; embolism protection; Carotid Stenosis
MeSH Terms: conditions — Stroke; Carotid Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAS with proximal protection (Experimental): using proximal embolism protection device during CAS
  Interventions: Device: proximal embolism protection device
- CAS with distal protection (Active Comparator): using distal protection device during CAS
  Interventions: Device: distal embolism protection device

INTERVENTIONS:
Device: proximal embolism protection device — a proximal occlusion Mo.Ma will be used as the embolism protection device during CAS
  Other Names: Mo.Ma Ultra (Invatec/Medtronic Vascular Inc, Santa Rosa, California)
  Arms: CAS with proximal protection
Device: distal embolism protection device — a distal SpiderFX will be used as the embolism protection device during CAS
  Other Names: SpiderFX (Medtronic, Minneapolis, Minnesota, USA)
  Arms: CAS with distal protection

SUMMARY:
A multicenter, prospective, outcome-assessor-blinded, randomized controlled trial study (MOSCASH) is designed to compare the efficiency of distal and proximal embolism protection devices during carotid angioplasty and stenting (CAS) procedure of patients with high-intensity signal in the plaque on the time-of-flight magnetic resonance angiography(TOF-MRA) .

DETAILED DESCRIPTION:
CAS is an alternative to carotid endarterectomy(CEA) for treating carotid stenosis with a similar efficacy in preventing future stroke. High-intensity signal in the plaque on the TOF-MRA is associated to a high risk of cerebral embolism during stenting. The evidence of protection selection in such patients was limited. A multicenter, prospective, outcome-assessor-blinded, randomized controlled trial study (MOSCASH) is designed to compare the efficiency of distal and proximal embolism protection devices during CAS procedure of patients with high-intensity signal in the plaque on the TOF-MRA. Asymptomatic patients with internal carotid artery stenosis ≥ 70% (NASCET) and symptomatic patients with a stenosis ≥ 50% who have a high-intensity signal in the relevant plaques on TOF-MRA will be included. Patients are randomized in two balanced groups (1:1) to receive CAS with either distal (Spider FX) or proximal (Mo.Ma Ultra) protection. The primary endpoint is the incidence of new cerebral ipsilateral ischemic lesions on the Diffusion Weighted Imaging(DWI) in 7-days post operation. Secondary endpoints include the number, size, location of new cerebral ischemic lesions on the DWI, procedural complications, stroke, myocardial infarction, and death in 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 40 years of age and older.
2. Asymptomatic patients with internal carotid artery stenosis≥70% on angiography.
3. Symptomatic patients with internal carotid artery stenosis≥50% on angiography.
4. High-intensity Signal in the relevant plaques on the TOF-MRA.
5. Anatomic characteristics of the lesions that made it possible to use either type of embolism protective device (proximal or distal).
6. The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent, approved by the appropriate Medical Ethics Committee, Institutional Review Board, or Human Research Ethics Committee.

Exclusion Criteria:

1. Extensive ipsilateral or disabling stroke(mRS≥2).
2. Ischemic ipsilateral stroke in 15 days, with significant new ischemic lesions on the DWI image.
3. Ipsilateral intracranial artery stenosis which needs to be treated at the same time.
4. Extremely calcified aortic arc that compromised the origin of the common carotid artery or the brachiocephalic trunk.
5. Chronic or paroxysmal atrial fibrillation treated with oral anticoagulation.
6. Acute coronary syndrome in the 30-day period before the procedure.
7. Patient has a history of bleeding diathesis within 1 month or coagulopathy or patients in whom antiplatelet and/or anticoagulant therapy is contraindicated.
8. Intolerance or allergic reaction to a study medication without a suitable management alternative.
9. Pregnant or lactating female patient.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
ipsilateral new ischemic lesions on DWI | within 7 days post-operation
  the incidence of ipsilateral new ischemic lesions on DWI after CAS

SECONDARY OUTCOMES:
major stroke | within 7 days post-operation
  the incidence of major stroke after CAS, defined as new onset of neurological symptoms causing an increase of NIHSS ≥ 4 or worsening of existing focal neurological deficit lasting ≥ 24 hours
myocardial infarction | within 7 days post-operation
  the incidence of myocardial infarction after CAS, defined as new onset of chest discomfort or cardiac stroke or heart failure with a rise and/or fall of cardiac biomarkers and ECG abnormalities
death | within 7 days post-operation
  In-hospital mortality
Other procedure-related complications | within 7 days post-operation
  including major/minor hemorrhage, acute kidney injury, etc.
The number, size, and location of new cerebral ischemic lesions on DW-MRI | within 7 days post-operation
  The number, size, and location of new cerebral ischemic lesions on DW-MRI

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Jiao, MD, PhD, Principal Investigator — Department of Neurosurgery & Interventional Neuroradiology Xuanwu Hospital
Locations (1):
- Xuanwu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data(IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: To share IPD in the magazine of paper published.

REFERENCES:
- [Background] Yoshimura S, Yamada K, Kawasaki M, Asano T, Kanematsu M, Takamatsu M, Hara A, Iwama T. High-intensity signal on time-of-flight magnetic resonance angiography indicates carotid plaques at high risk for cerebral embolism during stenting. Stroke. 2011 Nov;42(11):3132-7. doi: 10.1161/STROKEAHA.111.615708. Epub 2011 Aug 25. PMID 21868725
- [Background] Cano MN, Kambara AM, de Cano SJ, Pezzi Portela LA, Paes AT, Costa JR Jr, Abizaid AA, Moreira SM, Sousa AG, Sousa JE. Randomized comparison of distal and proximal cerebral protection during carotid artery stenting. JACC Cardiovasc Interv. 2013 Nov;6(11):1203-9. doi: 10.1016/j.jcin.2013.07.006. PMID 24262620
- [Background] Akkaya E, Vuruskan E, Gul ZB, Yildirim A, Pusuroglu H, Surgit O, Kalkan AK, Akgul O, Akgul GP, Gul M. Cerebral microemboli and neurocognitive change after carotid artery stenting with different embolic protection devices. Int J Cardiol. 2014 Sep 20;176(2):478-83. doi: 10.1016/j.ijcard.2014.07.241. Epub 2014 Aug 12. PMID 25125014